CLINICAL TRIAL: NCT02001844
Title: Single Blinded RCT to Investigate the Clinical Effectiveness of Pre-formed Semi-rigid Foot Orthoses (FOs) on Pain, Quality of Life and Dynamic of Gait With Children Diagnosed With Juvenile Idiopathic Arthritis (JIA).
Brief Title: Foot Orthoses (FOs) on Pain, Quality of Life and the Gait With Children Diagnosed With JIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Newcastle, Australia (Other)
Collaborators: Queen Margaret University (Other)
Responsible Party: Principal Investigator, Dr Andrea Coda, Dr, University of Newcastle, Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JIA - FOs intervention
Record Dates: First submitted 2013-11-25; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Arthritis, Juvenile Rheumatoid
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): The control FOs, or placebo FOs was supplied to patients who were randomly included in the control group. The control FOs was made of leather board (1mm), grey Poron (1mm), and black EVA (0.75mm) as covering. This thin inner sole did not have any sort of biomechanical support, nor had it any effect on the distribution of pressure, as it was completely flat. In addition, the placebo FOs did not present with any intrinsic or extrinsic correction underneath the sub-talar-joint (STJ).
  The use of black EVA as the covering material and the leather-board as a base, allowed for gathering of a dynamic impression over the 6 months of the trial.
  Interventions: Device: placebo foot orthoses (FOs)
- Trial Group (Experimental): Trial Group:
  children who were randomly introduced into this group received the pre-formed semi-rigid FOs. The FOs were used as an off the-shelf device and subsequently customised with chair side modifications. In order to reproduce the exact same aesthetical appearance as the control FOs, grey poron (1mm) and black EVA (0.75mm) was used as well to cover the trial FOs.
  Furthermore, depending on the type of correction applied to the trial patient, the black EVA also allowed the correction applied on the surface of the device to be masked.
  Interventions: Device: Trial Foot Orthoses (FOs)

INTERVENTIONS:
Device: Trial Foot Orthoses (FOs) — Trial Group:
  The children who were randomly introduced into this group received the pre-formed semi-rigid FOs. The FOs were used as an off the-shelf device and subsequently customised with chair side modifications. In order to reproduce the exact same aesthetical appearance as the control FOs, grey poron (1mm) and black EVA (0.75mm) was used as well to cover the trial FOs.
  Furthermore, depending on the type of correction applied to the trial patient, the black EVA also allowed the correction applied on the surface of the device to be masked.
  Arms: Trial Group
Device: placebo foot orthoses (FOs) — The control FOs, or placebo FOs was supplied to patients who were randomly included in the control group. The control FOs was made of leather board (1mm), grey Poron (1mm), and black EVA (0.75mm) as covering. This thin inner sole did not have any sort of biomechanical support, nor had it any effect on the distribution of pressure, as it was completely flat. In addition, the placebo FOs did not present with any intrinsic or extrinsic correction underneath the sub-talar-joint (STJ).
  The use of black EVA as the covering material and the leather-board as a base, allowed for gathering of a dynamic impression over the 6 months of the trial.
  Arms: Control

SUMMARY:
Modern modular foot-orthoses systems allow an integration of the cost and efficiency benefits afforded by the use of pre-formed semi-rigid FOs components, while simultaneously allowing a high degree of individualisation of prescription. Such systems, while popular, still remain unproven. Recent studies in paediatric rheumatology have made a contribution in developing guidelines with regards to pharmacological intervention in arthritic children. In addition, specific drug therapy protocols have been published to effectively help general practitioners, physiotherapists and ophthalmologists to successfully treat children with JIA patients (BSPAR 2006; Hull 2001; NICE guidelines 2002). A Cochrane systematic review on treatment of pes planus, highlighted that children with JIA were excluded as a group from most of the studies (Ashford et al. 2005). At present little evidence exists for the podiatric management of children affected by this disabling pathology, especially for orthotic management. This research has provided evidence to support the use of readily available off-the-shelf FOs in treating JIA children.

DETAILED DESCRIPTION:
Introduction - Currently there is limited evidence supporting podiatric treatment of children with JIA. The foot orthoses (FOs) prescribed to JIA children so far appeared to be very expensive and required long time to manufacture before the fitting. This randomised controlled trial (RCT) aimed to determine whether pre-formed FOs that can be prescribed at chair side, impacted on pain, quality of life (primary outcomes) and/or gait-parameters (secondary outcomes) in children affected by JIA.

Methods - The study took place at the Gait Analysis laboratory at Queen Margaret University - Edinburgh and at the TORT Centre, Ninewells Hospital-Dundee. Children with JIA were diagnosed according to the ILAR criteria. Intervention was blinded to the patients. The trial group received Slimflex-plus FOs, with the addition of chair side corrections and the control FOs supplied were made with leather board (1mm thick) only. Both FOs had the same black EVA top cover. Primary outcomes were investigated using validated questionnaires (VAS, CHAQ and PedsQL). Tekscan™ equipment (F-Scan™ and HR Walkway®) measured secondary outcomes in-shoe pressure and force data with and without FOs intervention. Multiple foot strikes and repetitive gait patterns were compared pre and post-treatment. Primary and secondary outcome measures were recorded at baseline, 3rd and 6th month's period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with JIA according to ILAR criteria.
* All subjects with lower extremity joint involvement with disease onset ranging from 5 to 18 years old.
* Previous failure of orthotic management, where the patient has not worn any FOs for a period of at least 3 months.
* Ability to walk a minimum of 15 metres without assistive devices.
* Six months after start of DMARD therapy.

Exclusion Criteria:

* Inability to walk barefoot or shod.
* Concomitant musculoskeletal disease, central or peripheral nerve disease and endocrine disorders, especially Diabetes Mellitus.
* Previous foot surgery.
* Currently using foot orthosis.
* Where supply of orthotics are contraindicated: (Less than 12 degrees at subtler joint; Fully compensated ankle equines; Osseous anomaly noted in the lower limbs and/or vertebrae during the physical evaluation; Inappropriate footwear for fitting orthoses).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
effects of pre-formed semi-rigid FOs on Pain in Paediatric Rheumatology. | 6 months
effects of pre-formed semi-rigid FOs on Quality of Life in Paediatric Rheumatology. | 6 months

SECONDARY OUTCOMES:
gait parameters when barefoot | 6 months
gait parameters with shoes | 6 months
gait parameters with shoes and foot orthoses (FOs) | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Dr Andrea Coda - Lecturer Podiatry , School of Health & Science, Ourimbah, New South Wales
  - University of Newcastle, Podiatry, School of Health & Science, Ourimbah, New South Wales

REFERENCES:
- [Derived] Coda A, Fowlie PW, Davidson JE, Walsh J, Carline T, Santos D. Foot orthoses in children with juvenile idiopathic arthritis: a randomised controlled trial. Arch Dis Child. 2014 Jul;99(7):649-51. doi: 10.1136/archdischild-2013-305166. Epub 2014 Mar 17. PMID 24636956